CLINICAL TRIAL: NCT05230810
Title: This is a Multicenter, Single Arm, Open-label, run-in Phase Ib / Roll-over Phase II Study of Tucatinib in Combination With Alpelisib in Subjects With PIK3CA-mutant HER2-positive Locally Advanced Unresectable or Metastatic Breast Cancer.
Brief Title: Clinical Trial of Alpelisb and Tucatinib in Patients With PIK3CA-Mutant HER2+ Metastatic Breast Cancer.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Criterium, Inc. (Industry)
Collaborators: Novartis (Industry); Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01AB21- PIK3CA
Record Dates: First submitted 2021-12-27; First posted 2022-02-09 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: HER2-positive Metastatic Breast Cancer
Keywords: ALPELISIB; TUCATINIB; HER2-positive Metastatic Breast Cancer
MeSH Terms: interventions — Alpelisib; tucatinib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ib Safety Cohort /II Expansion Cohort (Experimental): In phase Ib, the tolerability of tucatinib and alpelisib combination will be confirmed and maximum tolerated dose determined. Therapy will be administered in 28 day cycles of tucatinib 300 mg PO BID and alpelisib 250 mg PO daily (dose level 1). Treatment will continue until unacceptable toxicity, disease progression, withdrawal of consent, or study closure. Fulvestrant will also be administered in patients with HR+/HER2+ metastatic breast cancer. Once RP2D is determined, the study will be continued to phase II, and new patients will enroll at RP2D. All patients in phase IB part, who are remaining on study at the time of initiation of phase II, will be rolled over to phase II. At that time, their study drug doses will be modified as follows: (1) if a patient is on the drug doses lower than RP2D, doses will not be increased; (2) if a patient is on a higher doses compared to RP2D, doses of study drugs will be changed to RP2D.
  Interventions: Drug: Alpelisib; Drug: Tucatinib; Drug: Fulvestrant

INTERVENTIONS:
Drug: Alpelisib — Orally twice a day
  Other Names: Piqray
Drug: Tucatinib — Orally once a day
  Other Names: Tukysa
Drug: Fulvestrant — 500 mg intramuscularly into the buttocks slowly
  *Fulvestrant will be administered only in patients with HR+/HER2+ metastatic breast cancer
  Other Names: Faslodex,

SUMMARY:
Phase IB/II clinical trial of Alpelisb and Tucatinib in patients with PIK3CA-Mutant HER2-positive metastatic breast cancer.

DETAILED DESCRIPTION:
This study is a multicenter, single arm, open-label, run-in phase Ib safety cohort with immediate roll over to a phase II clinical trial that will test the combination therapy of tucatinib with alpelisib in subjects with PIK3CA-mutant HER2+ locally advanced unresectable or metastatic breast cancer. Patients with PIK3CA-mutant HR-/HER2+ and HR+/HER2+ breast cancer may enroll, the latter cohort will receive concomitant treatment with standard doses of fulvestrant to block HR signaling. In phase Ib part, we will confirm the tolerability of tucatinib and alpelisib combination and determine the maximum tolerated dose (MTD). In phase II part, we will expand the testing of this drug combination at MTD to determine the PFS rate.

ELIGIBILITY:
Criteria:

Inclusion criteria:

1. Women and men ≥ 18 years old are eligible to enroll
2. ECOG performance status 0-1
3. Life expectancy of more than 6 months, in the opinion of the investigator
4. Histologically confirmed diagnosis of HER2+ locally advanced unresectable or metastatic breast cancer. HER2 positivity is defined by fluorescence in situ hybridization (FISH) and/or 3+ staining by IHC according to the latest ASCO/CAP guidelines.
5. Documented presence of activating mutation in PIK3CA in the tumor, based on the analysis of solid or liquid biopsy by an assay approved for clinical decision makingby an FDA-approved test (examples include FoundationOne Liquid®; Guardant360®, Therrascreen® PIK3CA).
6. Known ER and PR status of the tumor defined by IHC according to the latest ASCO/CAP guidelines
7. Patients with HR-/HER2+ or HR+/HER2+ breast cancer may enroll
8. HR+/HER2+ patients should be men or post-menopausal women; premenopausal women with HR+/HER2+ breast cancer are eligible if on ovarian suppression, or agreeable to mandatory ovarian suppression
9. HR+/HER2+ patients should be agreeable to concomitant treatment with fulvestrant per study protocol. Prior therapy with fulvestrant is allowed.
10. Patients should have received at least two FDA-approved HER2-targeted agents at any time in the course of their disease. Note: 1 line of therapy containing EGFR or HER2-tyrosine kinase inhibitors (for example, neratinib, tucatinib, lapatinib, afatinib, pyrotinib, etc.) in the metastatic setting is allowed
11. Measurable and/or evaluable disease per RECIST 1.1 criteria and/or RANO-BM criteria (appendix C). Bone only disease is allowed.
12. CNS inclusion criteria:

Based on screening contrast brain MRI, patients must have one of the following:

1. No evidence of brain metastases 2. Untreated brain metastases not needing immediate local therapy. For patients with untreated CNS lesions > 2.0 cm on screening contrast brain MRI, discussion with and approval from the medical monitor is required prior to enrollment 3. Previously treated brain metastases

a. Brain metastases previously treated with local therapy may either be stable since treatment or may have progressed since prior local CNS therapy, provided that there is no clinical indication for immediate re-treatment with local therapy in the opinion of the investigator b. Patients treated with CNS local therapy for newly identified lesions found on contrast brain MRI performed during screening for this study may be eligible to enroll if all of the following criteria are met: i. Time since WBRT is ≥ 21 days prior to first dose of treatment, time since surgical resection of CNS metastases is ≥ 14 days prior to the first dose of study treatment, or time since SRS is ≥ 7 days prior to first dose of treatment.

ii. Other sites of disease evaluable by RECIST 1.1 or RANO-BM are present c. Relevant records of any CNS treatment must be available to allow for classification of target and non-target lesions. 13. Adequate organ and marrow function as defined below:

* Absolute neutrophil count ≥ 1,500/mm3
* Platelets ≥ 75,000/mm3
* Hemoglobin ≥ 9.0 mg/dL without red blood cell transfusion ≤ 7 days prior to Cycle 1 Day 1 of therapy
* Total serum bilirubin ≤ 1.5 X upper limit of normal (ULN) except for subjects with known Gilbert's disease, who may enroll if the conjugated bilirubin is ≤ 1.5 ULN
* AST (SGOT)/ALT (SGPT) ≤2.5 X ULN;
* Serum creatinine Estimated creatinine clearance ≥50 mL/min as calculated by Cockroft-Gault formula; actual body weight must be used for creatinine clearance calculations unless BMI > 30 kg/m2 then lean body weight must be used;≤ 1.5 mg/dL
* International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 X ULN unless on medication known to alter INR and aPTT
* Fasting blood glucose ≤140 mg/dL
* HbA1C≤6.4%
* Left ventricular ejection fraction (LVEF) ≥ 50% (as assessed by ECHO or MUGA) documented within 4 weeks prior to first dose of study treatment
* Serum or urine pregnancy test (for women of childbearing potential, defined as premenopausal women who are not permanently sterile due to hysterectomy, bilateral oophorectomy, bilateral tubal ligation, or bilateral tubal occlusion) negative ≤ 7 days of starting treatment 14. Patients with body mass index >25, or FBG 110-140mg/dL, or HbA1C 5.7 - 6.4% should be agreeable for low glycemic diet and lifestyle modifications, and consulted by nutritionist prior to initiation of the study drugs. Ability to understand and the willingness to sign a written informed consent and comply with the study scheduled visits, treatment plans, laboratory tests and other procedures.

Exclusion criteria:

1. Patients with contraindications to undergo contrast MRI imaging of the brain are excluded from the study
2. Pregnancy or breast feeding
3. Any systemic anti-cancer therapy (including hormonal therapy or investigational agents) or surgery in <14 days prior to the first dose of study treatment WBRT in <21 days, SBRT for CNS disease in <7 days, or palliative radiation to extracranial sites in <14 days prior to the first dose of study treatment5.
4. Based on screening brain MRI, patients must not have any of the following:

1. Any untreated brain lesions > 2.0 cm in size, unless discussed with medical monitor and approval for enrollment is given 2. Ongoing use of systemic corticosteroids for control of symptoms of brain metastases at a total daily dose of > 2 mg of dexamethasone (or equivalent). However, patients on a chronic stable dose of ≤ 2 mg total daily of dexamethasone (or equivalent) may be eligible with discussion and approval by the medical monitor 3. Any brain lesion thought to require immediate local therapy, including (but not limited to) a lesion in an anatomic site where increase in size or possible treatment-related edema may pose risk to patient (e.g. brain stem lesions). Patients who undergo local treatment for such lesions identified by screening contrast brain MRI may still be eligible for the study based on criteria described under CNS inclusion criteria 3b 4. Known or suspected leptomeningeal disease as documented by the investigator 5. Have poorly controlled (> 1/week) generalized or complex partial seizures, or manifest neurologic progression due to brain metastases notwithstanding CNS-directed therapy 5. Any toxicity related to prior cancer therapies that has not resolved to ≤ Grade 1, with the exception of peripheral neuropathy, which must have resolved to ≤ Grade 2, and alopecia 6. More than 1 line of therapy containing tucatinib, lapatinib, neratinib, afatinib, pyrotinib, or other EGFR or HER2 tyrosine kinase inhibitor in the metastatic setting. Note: receiving the above medications for <30 days is not considered to be a "line of therapy". Adjuvant treatment with EGFR or HER2 tyrosine kinase inhibitors does not count.

7. Previous treatment with alpelisib or other PI3K, mTOR or AKT inhibitor of more than 30 days duration.

8. An established diagnosis of diabetes mellitus type I, or uncontrolled diabetes mellitus type II 9. History of acute pancreatitis within 1 year of screening, or a past medical history of chronic pancreatitis 10. History of severe cutaneous hypersensitivity reactions (Steven Johnson syndrome, erythema multiforme or toxic epidermal necrolysis) 11. Active bacterial, fungal or viral infections requiring treatment with IV antibiotic, IV anti-fungal, or IV anti-viral drugs 12. Known active hepatitis B (HBV) or, active hepatitis C (HCV) or human immunodeficiency virus (HIV) infections. Note: pretesting is not required. Patients with history of treated and cured HCV infection may enroll if they have documented undetectable viral load.

13. Known HIV infection with CD4+ T-cell (CD4+) counts < 350 cells/μL. Note: pretesting is not required. Patients with known HIV infection and CD4+ T-cell (CD4+) counts ≥ 350 cells/μL may enroll.

14. Inability to swallow pills or any significant gastrointestinal disease which would preclude the adequate oral absorption of medications 15. Use of prohibited medications listed in the Appendix D (strong CYP3A4 inducers or inhibitors, and strong CYP2C8 inducers or inhibitors) within 3 elimination half-lives prior to initiation of study treatments 16. Myocardial infarction, severe/unstable angina, percutaneous transluminal coronary angioplasty/stenting (PTCA), or coronary artery bypass graft (CABG) within 6 month of the first dose of the study treatment 17. Clinically significant cardio-vascular disease, such as ventricular arrhythmia requiring therapy, uncontrolled hypertension (defined as persistent systolic blood pressure > 160 mm Hg and/or diastolic blood pressure > 100 mm Hg on antihypertensive medications), or any history of symptomatic congestive heart failure (CHF) 18. Other severe acute or chronic medical or psychiatric conditions or laboratory abnormalities that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, or in the judgment of the investigator would make the subject inappropriate for entry into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-08-25 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Phase Ib Safety and Tolerability of alpelisib and tucatinib combination, summary of all AEs and SAEs on study as evaluated by NCI-CTCAE v 5.0 | 10 Months
  MTD of tucatinib and alpelisib in combination, summary of all AEs and SAEs on study as evaluated by NCI-CTCAE v 5.0
Phase II Efficacy of tucatinib combination evaluated by progression free survival (PFS) | 20 Months
  PFS in the overall study population (the time from allocation to the first documented disease progression by RECIST1.1, or death due to any cause, whichever occurs first)

SECONDARY OUTCOMES:
Phase Ib Pharmacokinetic (PK) properties of alpelisib and tucatinib | 10 Months
  Plasma concentrations of alpelisib and tucatinib measured at cycle 1 day 15 of therapy
Phase Ib Tumor response evaluation | 10 Months
  CR, PR, or SD according to RECIST 1.1 (for subjects with CNS disease by RECIST 1.1 and RANO-BM); assessment of ORR (CR and PR), CBR (CR, PR and SD)
Phase Ib Duration of Response (DOR) | 10 months
  Duration of response defined as the time from enrollment into clinical trial until objective tumor progression or death whichever occurs first.
Phase II Tumor response evaluation | 20 months
  CR, PR, or SD according to RECIST 1.1 (for subjects with CNS disease by RECIST 1.1 and RANO-BM); assessment of ORR (CR and PR), CBR (CR, PR and SD)
Phase II Incidence, nature and severity of all AEs that occur on or after C1D1 of therapy | 20 months
  Safety and tolerability of the combination therapy
Phase II Duration of Reponse (DOR) | 20 months
  duration of response (DOR) defined as the time from enrollment into clinical trial until objective tumor progression or death whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Shagisultanova, MD, Principal Investigator — University of Colorado, Denver
Locations (4):
- United States (4):
  - University of Colorado Cancer Center, Aurora, Colorado
  - Cancer Care & Hematology-Fort Collins, Fort Collins, Colorado
  - Louisiana State University Health Sciences Center, New Orleans, Louisiana
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin